CLINICAL TRIAL: NCT00213902
Title: Evaluation of Effects of Central Sympathetic Inhibition in Elderly With Left Ventricular Diastolic Dysfunction and Preserved Ejection Fraction: A Proof-of-Concept Trial With Clonidine
Brief Title: Clonidine and Left Ventricular Dysfunction
Status: Withdrawn | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Other Study IDs: 3153
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Ventricular Dysfunction
Keywords: Heart failure; Diastolic; functionClonidine; Left ventricular diastolic dysfunction with preserved ejection fraction
MeSH Terms: conditions — Ventricular Dysfunction; Heart Failure; Heart Murmurs

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The objectives of this study are:

1. To evaluate the effect of clonidine, a sympathetic modulator, to reverse cardiac remodeling and to improve hemodynamics in diastolic heart failure (DHF).
2. To evaluate the effect of clonidine on neurohormones and quality of life in patients with DHF.

The study is a double-blind, placebo-controlled study evaluating the effects of clonidine compared to placebo in patients with DHF. A total of 70 patients with DHF will be randomized in a 1:1 ratio to:

1. placebo (n=35) or to
2. clonidine (n=35) in a dose of 0.075 mg twice a day for the first 6 weeks followed by uptitration to 0.150 mg twice a day for 6 months.

The primary outcome is the reversion of cardiac remodeling and hemodynamic parameters evaluated by magnetic resonance imaging (MRI) and echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60 and greater
* Gender: Both
* Patients with heart failure New York Heart Association (NYHA) II and ejection fraction over 45%

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Bousquet, MD, Principal Investigator — Hopitaux Universitaires de Strasbourg